CLINICAL TRIAL: NCT05974345
Title: In Silico Non Interventional Secondary Use of Data Study Assessing the Impact of Inclisiran on Major Adverse Cardiovascular Events in Patients With Established Cardiovascular Disease
Brief Title: In Silico Study Assessing the Impact of Inclisiran on Major Adverse Cardiovascular Events in Patients With Established Cardiovascular Disease
Acronym: SIRIUS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839B1FR01
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Atherosclerotic cardiovascular disease; Hypercholesterolemia; Dyslipidemia; High cholesterol; Hyperlipidemia; Inclisiran; siRNA; KJX839; Myocardial infarction; Ischemic stroke; Peripheral arterial disease; In silico model; In silico simulation; PCSK9 inhibitors; Arteriosclerosis; Atherosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Dyslipidemias; Hyperlipidemias; Myocardial Infarction; Ischemic Stroke; Peripheral Arterial Disease; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Ezetimibe; evolocumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual Patient with ASCVD: Virtual Patient with ASCVD and LDL-C ≥ 70 mg/dL despite receiving a well-tolerated high-intensity statin with or without ezetimibe. Each virtual patient is his own control.
  Interventions: Drug: Inclisiran sodium; Drug: Placebo; Drug: Ezetimibe; Drug: Evolocumab

INTERVENTIONS:
Drug: Inclisiran sodium — Drug: Inclisiran sodium 300 mg virtually subcutaneously administered on Day 1, Month 3 (Day 90) and every 6 months thereafter until end of simulation.
Drug: Placebo — Drug: Placebo virtually subcutaneously administered on Day 1, Month 3 (Day 90) and every 6 months thereafter until end of simulation.
Drug: Ezetimibe — Drug: Ezetimibe 10 mg virtually orally once a day until end of simulation.
Drug: Evolocumab — Drug: Evolocumab 140 mg virtually subcutaneously administered every two weeks until end of simulation.

SUMMARY:
Study CKJX839B1FR01 in an In silico trial to predict the efficacy of Inclisiran therapy on major adverse cardiovascular events (MACE) and cardiovascular (CV) death in virtual patients with atherosclerotic cardiovascular disease (ASCVD) and elevated LDL-C.

DETAILED DESCRIPTION:
Purpose of this study is to predict the size of efficacy of inclisiran 300 mg s.c., administered on Day 1, Month 3 (Day 90), and every 6 months thereafter in addition to currently available lipid lowering therapies (LLTs) on a 3-Point-Major Adverse Cardiovascular Events (3P-MACE) defined as a composite of CV death, non-fatal myocardial infarction (MI) or non-fatal ischemic stroke, and on CV death, in a secondary prevention cohort of ASCVD virtual patients with a LDL-C ≥ 70 mg/dL. This will be compared to 1) placebo in adjunct to high-intensity statin therapy with or without ezetimibe, 2) ezetimibe in adjunct to high-intensity statin therapy, 3) Evolocumab in adjunct to high-intensity statin therapy and ezetimibe.

ELIGIBILITY:
Inclusion Criteria :

1. Patients with atherosclerotic CV disease, defined as any of the following

   i. Previous MI

   ii. Previous ischemic stroke

   iii. Previous symptomatic peripheral arterial disease (PAD) as evidenced by either intermittent claudication with ABI <0.85, prior peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease
2. Fasting LDL-C ≥ 70 mg/dL
3. Under stable (≥ 4 weeks) well-tolerated high-intensity statin with or without ezetimibe.

Exclusion Criteria :

Patients with acute coronary syndrome, ischemic stroke, peripheral arterial revascularization procedure or amputation due to atherosclerotic disease <4 weeks prior to the first study visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Virtual Patient with ASCVD (previous MI, previous ischemic stroke, previous peripheral arterial disease) and LDL-C ≥ 70 mg/dL despite receiving a well-tolerated high-intensity statin with or without ezetimibe.
Sampling Method: Non-Probability Sample
Enrollment: 204691 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Time to the first occurrence between trial start and end of follow-up of any component of 3P-MACE (composite of CV death, non-fatal MI or non-fatal ischemic stroke) | 5 years of follow-up
  3P-MACE is a confirmed composite endpoint which includes cardiovascular death, non-fatal myocardial infarction and non-fatal ischemic stroke.
Time to the first occurrence between trial start and end of follow-up of CV death | 5 years of follow-up
  CV death is defined as death due to cardiovascular events

SECONDARY OUTCOMES:
Time to the first occurrence between trial start and end of follow-up of MI (non-fatal or fatal) | 5 years of follow-up
  Myocardial infarction (MI)
Time to the first occurrence between trial start and end of follow-up of ischemic stroke (non-fatal or fatal) | 5 years of follow-up
Time to the first occurrence between trial start and end of follow-up of Major Adverse Limb events (MALE) | 5 years of follow-up
  MALE include acute lower limb ischemia, lower limb amputation due to ischemia, or urgent lower limb revascularization for ischemia
Change in LDL-C from baseline to specified time points | baseline, day 1, 30, 90 and every 6 months afterwards will be presented and additional time points could be added if deemed necessary.
  Low density lipoprotein cholesterol (LDL-C)
Time adjusted percentage change in LDL-C | From baseline between Day 90 and the end of follow-up period (up to 5 years)
  This is the average percentage change in LDL-C from baseline over period from Day 90 and the end of follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Rueil-Malmaison, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angoulvant D, Granjeon-Noriot S, Amarenco P, Bastien A, Bechet E, Boccara F, Boissel JP, Cariou B, Courcelles E, Diatchenko A, Filipovics A, Kahoul R, Mahe G, Peyronnet E, Portal L, Porte S, Wang Y, Steg PG. In-silico trial emulation to predict the cardiovascular protection of new lipid-lowering drugs: an illustration through the design of the SIRIUS programme. Eur J Prev Cardiol. 2024 Nov 11;31(15):1820-1830. doi: 10.1093/eurjpc/zwae254. PMID 39101472